CLINICAL TRIAL: NCT06436937
Title: Protein Quality of Fava Bean Meat Analogue and Honey Chlorella Ingested as Mixed Meals in Healthy Volunteers
Brief Title: Protein Quality of Fava Bean and Honey Chlorella in Humans
Acronym: Giant Leaps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor in Gastroenterology, Assistance Publique - Hôpitaux de Paris
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GIANT LEAPS
Record Dates: First submitted 2024-04-10; First posted 2024-05-31 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Protein Quality of Chlorella and Fababean Meat Analogue
Keywords: Digestibility; healthy humans; nasoileal tubes; stable isotopes; nitrogen retention; postprandial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey Chlorella (Experimental): The subjects ingest a single meal: a drink including 40 g of honey chlorella intrinsically labelled with 15N, to provide 20g protein from chlorella
  Interventions: Dietary Supplement: Single meal containing 20 g of 15N intrinsically labelled protein from honey chlorella
- Faba bean meat analogue (Experimental): The subjects ingest a single meal: a mixed meal including 80 g of faba bean meat analogue intrinsically labelled with 15N, to provide 20g protein from faba bean
  Interventions: Dietary Supplement: Single meal containing 20 g of 15N intrinsically labelled protein from faba bean meat analogue

INTERVENTIONS:
Dietary Supplement: Single meal containing 20 g of 15N intrinsically labelled protein from honey chlorella — Ingestion of a 15N labeled test meal. Subjects are equipped with a nasoileal tube. 15N is followed in biological fluids (plasma, effluents, urines).
  Arms: Honey Chlorella
Dietary Supplement: Single meal containing 20 g of 15N intrinsically labelled protein from faba bean meat analogue — Ingestion of a 15N labeled test meal. Subjects are equipped with a nasoileal tube. 15N is followed in biological fluids (plasma, effluents, urines).
  Arms: Faba bean meat analogue

SUMMARY:
The goal of the project is to determine the protein quality of alternative protein sources, honey chlorella and Faba bean, ingested as mixed meals in healthy subjects equipped with naso-ileal tube. For this purpose, Chlorella and Faba bean are intrinsically labelled with 15N. Faba bean is processed to produce a meat analogue. Chlorella is introduced in a drink. The protein quality is determined by following the digestive and metabolic fate of 15N during a 8h postprandial investigation.

DETAILED DESCRIPTION:
The objective is to determine the nutritional quality of protein from honey chlorella and faba bean meat analogue in healthy humans, especially in terms of protein and amino acid digestibility as well as nitrogen retention. Ileal digestibility is determined in ileal digesta collected postprandially with a naso-ileal tube. The protein sources are intrinsically labelled in 15N in order to track dietary nitrogen and amino acids in the samples.

Ethical and regulatory aspects:

The protocol has been approved to the Ethical Committee and authorized the French Agency of Drugs and Health. The personal data management will be in accordance with the regulation on personal data protection ( " regulation n° 2018-493 du 20 juin 2018").

Meal:

The meal will consist in either a drink containing 40 g of honey chlorella or a mixed meal containiong 80 g of meat analogue, to provide 20 g protein. Sensory tests will be realized to optimize the organoleptic properties of the meal.

Volunteers:

Sixteen subjects will be included in the study. The investigators plan to recruit around 40 volunteers to accommodate for the usual 60% dropouts.

Four days before the experiment, the volunteers will follow a standard diet adapted to their body weight to control their protein intake (1.3 g protein/kg body weight).

The volunteers will arrive at the Human Nutrition Research Centre of Avicenne Hospital on the morning before the day of the experiment. They will be equipped with a double lumen intestinal tube that will be allowed to progress through the intestinal tract for 24h. One of the lumen is radio opaque and serves to perfuse a non-absorbable maker in the intestine (slow marker method). The other lumen is dedicated to the continuous aspiration of the effluents, 15 cm below the perfusion site. The measurement of the non-absorbable marker in the effluents allows the determination of the effluent flow rate.

On the evening before the experimental day, they will ingest 3 oral doses of deuterated water 99 % to reach 5g/kg total body water, to label the intestinal endogenous proteins.

On the day of the experiment, the position of the tube will be checked by radiography to verify its location at the terminal ileum. A catheter will be inserted in the forearm vein for blood sampling. The perfusion of the non-absorbable marker, PEG-4000 (20g/l), will start at a flow rate of 1ml/min. The intestinal flow and the basal ileal sample will be collected during 30 min. Basal plasma sample will be sampled.

Then, at t=0, the volunteers will drink the test-meal. Until t=8h, intestinal content will be continuously collected by aspiration and pooled every 30 minutes. Blood will be sampled every 30 minutes during 4h and hourly thereafter. The urine will be collected every 2 h for 8 h.

Measurements:

In the ilel digesta:

PEG-4000 by turbidimetric method, total N and 15N enrichment by EA-IRMS, amino acid concentrations by UPLC (after acid hydrolysis HCl 6N at 110°C for 24h), 15N amino acid enrichment by GC-c-IRMS (after purification on cation exchange resin and derivatization), 2H amino acid enrichment by GC-c-IRMS, microbiome analysis (DNA sequencing), peptide analysis (LC-MS).

In the plasma:

Glucose, urea (colorimetric methods), insulin (ELISA), amino acid concentrations (UPLC), 15N enrichment in plasma protein, urea and free amino acids (EA-IRMS, after purification on cation exchange resin and derivatization).

In the urine:

Urea (colorimetric method) and 15N urea (EA-IRMS, after purification on cation exchange resin and derivatization).

Main outcomes are:

Real ileal digestibility of protein and amino acids (digestive losses), Postprandial deamination (metabolic losses), Net Postprandial Protein Utilization

ELIGIBILITY:
Inclusion Criteria:

* 18<BMI<30
* Good health (WHO=0)
* For woman: use of birth control

Exclusion Criteria:

* food allergy
* allergy against latex
* pregnant women
* Positive serology for AgHBS, AcHbc, HCV, HIV
* Anemia
* Excessive alcohool consumption
* Hypertension, diabetes, digestive, hepatic or renal diseases, cardiac disease
* Exercice>7h/week
* Blood donation within 3 months before the study
* Participation to another clinical study within 3 months before the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Ileal digestibility of protein and amino acids | -30 minutes to 8 hours after the test meal
  The measurement of nitrogen (mmol) and 15N enrichment (atom %) in ileal samples allow to determine the amount of dietary nitrogen in the lumen. Dietary nitrogen that is recovered in the ileal samples are then considered as non absorbed.
Net Postprandial Protein Utilization (NPPU) | 0 to 8 hours after the test meal
  The measurement of urea (mmol) and 15N enrichment of urea (atom %) allow to determine the amount of dietary N that was transferred to urea, thus accounting for metabolic losses. Metabolic losses of dietary N, together with digestive losses of dietary N, are not retained in the body.
Ileal digestibility of amino acids | -30 minutes to 8 hours after the test meal
  The measurement of amino acid concentration (mmol) and their individual 15N enrichment (atom %) allow the determination of dietary amino acids remaining in the lumen. Dietary amino acids that are recovered in the ileal samples are then considered as non absorbed.

SECONDARY OUTCOMES:
Nitrogen metabolites in blood in response to the ingestion of 15N fava bean | 0 to 8 hours after the test meal
  urea and amino acids (mmol/l)
Plasma glucose in blood in response to the ingestion of 15N fava bean | 0 to 8 hours after the test meal
  plasma glucose (mmol/l)
Plasma insulin in blood in response to the ingestion of 15N fava bean | 0 to 8 hours after the test meal
  plasma insulin (pmol/l)
Ileal microbiota | -0.5 h before the meal
  Microbial DNA sequencing
Peptide composition of ileal digesta | 0-8 h after the test meal
  Peptidomic anlaysis by LC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Claire Gaudichon, PhD, Prof, Study Director — INRAE; Robert Benamouzig, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Research Center on Volunteers, Bobigny, France